CLINICAL TRIAL: NCT05142917
Title: The Effect of tDCS Based on Functional Brain Imaging for Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-10-092-001
Record Dates: First submitted 2021-11-28; First posted 2021-12-03 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2021-11

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fNIRS based hand motor area real stimulation (Experimental): Real stimulation is applied to functional brain image-based hand function area (20 minutes) and then hand motor task (20 minutes).
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Hand motor task
- Traditional hand motor area real stimulation (Active Comparator): Real stimulation is applied to the traditional hand function area (20 minutes) and then hand motor task (20 minutes).
  Interventions: Device: Transcranial Direct Current Stimulation; Behavioral: Hand motor task
- Traditional hand motor area sham stimulation (Sham Comparator): Sham stimulation is applied to the traditional hand function area (20 minutes) and then hand motor task (20 minutes).
  Interventions: Behavioral: Hand motor task

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial direct current stimulation is a form of noninvasive neuromodulation that uses constant and low direct current delivered via electrodes on the scalp.
  Arms: Traditional hand motor area real stimulation; fNIRS based hand motor area real stimulation
Behavioral: Hand motor task — Various type of hand motor tasks are applied to stroke patients.

SUMMARY:
The purpose of this study is to investigate whether brain imaging-based hand function area tDCS stimulation is more effective than conventional stimulation or sham stimulation for improving hand motor function.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral stroke patients aged 19 to 80 years
* Patients with subacute stroke within 4 weeks of onset
* Patients with moderate or severe upper extremity dysfunction with an upper extremity FMA score of less than 58 in motor function evaluation

Exclusion Criteria:

* Accompanied by an existing serious neurogenic disease
* Existing significant psychiatric disorders such as major schizophrenia, bipolar disorder, and dementia.
* If there are difficulties in conducting the research
* Any patients who are judged by the investigator to be difficult to participate in this study
* Exclusion criteria for transcranial direct current stimulation:

  i) Patients with implanted medical devices in the body (e.g. pacemakers) ii) When a metal object is inserted in the skull iii) If there is a wound on the skin of the attachment site iv) history of epilepsy v) Pregnant and lactating women

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-01-08 (Actual)

PRIMARY OUTCOMES:
Changes of score: Fugl-Meyer Assessment | Baseline, within 48 hours after #1-10 brain stimulation sessions (5 times per week, total 2 week schedule), 1 month after ten brain stimulation session
  The score is a stroke-specific, performance-based impairment index. The degree of impairment of upper and lower limbs is measured.

SECONDARY OUTCOMES:
Changes of score: 9-hole pegboard test | Baseline, within 48 hours after #1-10 brain stimulation sessions (5 times per week, total 2 week schedule), 1 month after ten brain stimulation session
  The test is a standardized, quantitative assessment used to measure finger dexterity of a patient.
Changes of score: Grip & Tip pinch strength test | Baseline, within 48 hours after #1-10 brain stimulation sessions (5 times per week, total 2 week schedule), 1 month after ten brain stimulation session
  The test is to measure the maximum isometric strength of hand, forearm, and finger muscles.
Changes in Box & Block test | Baseline, within 48 hours after #1-10 brain stimulation sessions (5 times per week, total 2 week schedule), 1 month after ten brain stimulation session
  The test is used to measure the gross manual dexterity of a patient, or of a person using an upper limb prosthetic device.
Changes of score: Jebsen-Taylor hand function test | Baseline, within 48 hours after #1-10 brain stimulation sessions (5 times per week, total 2 week schedule), 1 month after ten brain stimulation session
  This test is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living (ADL).
Changes of score: Korean-Montreal Cognitive Assessment | Baseline, within 48 hours after #1-10 brain stimulation sessions (5 times per week, total 2 week schedule), 1 month after ten brain stimulation session
  This test is a cognitive function test tool consisting of spatiotemporal/executive function, naming, memory, attention, language function, abstraction, and orientation.
Changes of score: Korean version of Modified Barthel Index | Baseline, within 48 hours after #1-10 brain stimulation sessions (5 times per week, total 2 week schedule), 1 month after ten brain stimulation session
  Measure of physical disability used widely to assess behaviour relating to activities of daily living for stroke patients or patients with other disabling conditions.
Changes of score: Geriatric Depression Scale-Short Form | Baseline, within 48 hours after #1-10 brain stimulation sessions (5 times per week, total 2 week schedule), 1 month after ten brain stimulation session
  The test is a self-report measure of depression in older adults.
Changes in cortical activity using fNIRS signals | Baseline, within 48 hours after #1-10 brain stimulation sessions (5 times per week, total 2 week schedule), 1 month after ten brain stimulation session
  Cortical activities before, during and after brain stimulation sessions are compared.

OTHER OUTCOMES:
Resting-state functional MRI | Baseline (Before stimulation sessions)
  Before intervention, MRI is acquired to extract brain characteristics of stroke patients.
Changes in cortical activity using fNIRS signals | Baseline (Before stimulation sessions)
  Before intervention, fNIRS image is acquired to extract cortical activation of stroke patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea